CLINICAL TRIAL: NCT00293917
Title: A Phase 3, Long-Term, Open Label Study to Evaluate the Safety of Twice Daily Tacrolimus Cream-B 0.1% in the Treatment of Psoriasis
Brief Title: A Study to Assess the Long-Term Safety of Tacrolimus Cream in the Treatment of Psoriasis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Collaborators: Astellas Pharma US, Inc. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 04-0-207
Record Dates: First submitted 2006-02-16; First posted 2006-02-20 (Estimated); Last update posted 2008-02-13 (Estimated); Status verified 2008-02

CONDITIONS: Psoriasis
Keywords: Treatment Outcome; Tacrolimus; Safety; Psoriasis
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Tacrolimus Cream

SUMMARY:
A study to assess the long-term safety of tacrolimus cream in the treatment of psoriasis

DETAILED DESCRIPTION:
A long-term, open label, non-comparative, multi-center study to evaluate the safety of tacrolimus cream-B 0.1% in treating the signs and symptoms of psoriasis.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of plaque psoriasis

Exclusion Criteria:

* Skin disorder other than plaque psoriasis in the areas to be treated.
* Disease on only scalp

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 658 (Actual)
Dates: Start 2006-01; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Safety | 12 months

SECONDARY OUTCOMES:
Efficacy | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: M Rico, MD, Study Director — Astellas Pharma US, Inc.
Locations (35):
- United States (29):
  - Birmingham, Alabama
  - Fresno, California
  - Santa Monica, California
  - Vista, California
  - Jacksonville, Florida
  - Miami, Florida
  - Atlanta, Georgia
  - Newnan, Georgia
  - Boise, Idaho
  - Chicago, Illinois
  - Louisville, Kentucky
  - New Orleans, Louisiana
  - Boston, Massachusetts
  - Detroit, Michigan
  - Minneapolis, Minnesota
  - Lincoln, Nebraska
  - Reno, Nevada
  - Lebanon, New Hampshire
  - East Windsor, New Jersey
  - East Setauket, New York
  - New York, New York
  - Hershey, Pennsylvania
  - Simpsonville, South Carolina
  - Goodlettsville, Tennessee
  - Arlington, Texas
  - Houston, Texas
  - Bellingham, Washington
  - Kenatchee, Washington
  - Spokane, Washington
- Canada (6):
  - Winnipeg, Manitoba
  - St. John's, Newfoundland and Labrador
  - Halifax, Nova Scotia
  - Hamilton, Ontario
  - Markham, Ontario
  - Windsor, Ontario